CLINICAL TRIAL: NCT00432120
Title: Clopidogrel Loading Dose for ad-Hoc Percutaneous Coronary Intervention Immediately Following Elective Coronary Angiography: Randomized Multicenter Trial Comparing Pre-Treatment > 6 Hours Before Every Angiography vs. Cath-Lab Administration After Angiography (Just Before Intervention): the PRAGUE-8 Trial.
Brief Title: Clopidogrel Only Before Percutaneous Coronary Intervention or Before Every Coronarography?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PRAGUE 8
Record Dates: First submitted 2007-02-05; First posted 2007-02-07 (Estimated); Last update posted 2008-01-29 (Estimated); Status verified 2007-08

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia | interventions — Clopidogrel

ARMS (2):
- A (Active Comparator): "nonselective" - clopidogrel 600 mg >6 hours before coronary angiography;
  Interventions: Drug: clopidogrel
- B (Active Comparator): "selective" - clopidogrel 600 mg in the cath-lab after coronary angiography, only in case of percutaneous coronary intervention
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: clopidogrel — To compare two different clopidogrel regimens on the outcomes of patients undergoing elective coronary angiography ± ad-hoc percutaneous coronary intervention

SUMMARY:
Clopidogrel pre-treatment before planned percutaneous coronary intervention was proved to reduce periprocedural complications. However, the vast majority of patients in the current interventional cardiology practice do not undergo planned PCI, but rather "ad-hoc" PCI performed immediately after coronary angiography . Whether clopidogrel should be administered as pre-treatment to all patients undergoing elective CAG with the aim to ensure therapeutic levels at the time of possible ad-hoc PCI is not known.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Elective CAG for suspected or proven coronary artery disease (stable forms or fully stabilized acute coronary syndrome)
3. Signed written informed consent

Exclusion Criteria:

1. Thienopyridine treatment in previous two weeks
2. Contraindication for clopidogrel
3. CAG scheduled less than 6 hours after potential randomization
4. Clinically significant bleeding (i.e. with hemoglobin fall by > 50 g/l and/or requiring transfusions or surgery) in previous 3 months.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2006-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Primary end point was the first clinical occurrence of any of the following: death / periprocedural myocardial infarction / stroke or transient ischemic attack / re-intervention | within 7 days

SECONDARY OUTCOMES:
Secondary end-points were periprocedural troponin elevation (> 3x ULN), TIMI-flow after PCI, bleeding complications and each individual component of the combined primary endpoint | within 7 day

CONTACTS AND LOCATIONS:
Overall Officials: Petr Widimsky, MD, Principal Investigator — Charles University, Prague, Czech Republic; Zuzana Motovska, MD, Principal Investigator — Charles University, Prague, Czech Republic
Locations (1):
- Charles University, Prague, Czechia